CLINICAL TRIAL: NCT02461498
Title: The AHEAD Study: Monitoring Anticoagulated Patients Who Suffer Head Injury
Status: Completed | Type: Observational
Sponsor: University of Sheffield (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Professor Suzanne Mason, Professor of Emergency Medicine, University of Sheffield
Other Study IDs: PB-PG-0808-17148
Record Dates: First submitted 2015-05-27; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Craniocerebral Trauma; Head Injuries, Closed
Keywords: Warfarin
MeSH Terms: conditions — Craniocerebral Trauma; Head Injuries, Closed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Existing practice in emergency departments (ED) in the United Kingdom (UK) for managing patients taking warfarin after a blunt head injury is variable with little research that supports the most appropriate way to manage these patients. The investigators aimed to undertake research in order to understand the range and frequency of outcomes following head injury in this group of patients and to develop robust clinical guidance for how they should be optimally managed in the future.

DETAILED DESCRIPTION:
This prospective observational study aims to enrol patients taking warfarin that attend participating ED's (up to 33) in England and Scotland after blunt head injury. Over an 18-month period from Oct 2011, ED attendance data will be collected from each ED as well as information from patient questionnaires about the care the patient received and the status of their health 6-10 weeks after the injury. Patients who died due to their head injury, experienced surgery due to their injury, had a change identified on a CT scan or re-attended the ED with a clear head injury complication are defined as experiencing a poor outcome. Information such as the patients' conscious state (GCS), level of clotting in their blood (INR) and symptoms will be investigated as predictors of a poor outcome. A mathematical model will be used to estimate the most cost-effective strategy assuming published National Institute for Health and Care Excellence (NICE) thresholds for cost per quality adjusted life year (QALY).

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older
* Blunt head trauma above the neck within 24 hours of ED attendance
* Prescribed warfarin

Exclusion Criteria:

* Penetrating injuries to the head, for example knife wound.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults who attend participating emergency departments (ED) with a head injury and also prescribed warfarin
Sampling Method: Non-Probability Sample
Enrollment: 3556 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Rate of head injury complication in study cohort | 18 months
  Head injury complications defined as death or neurosurgery resulting from the initial injury, a clinically-significant CT scan finding or re-attendance to the ED with a significant head injury-related complication up to 10 weeks after the original attendance.

SECONDARY OUTCOMES:
Prevalence of ongoing symptoms relating to the head injury | 18 months
  Impaired activities of daily living (assessed by the EQ5D)
Prevalence of ongoing symptoms relating to the head injury | 18 months
  Headache symptoms
Prevalence of ongoing symptoms relating to the head injury | 18 months
  Impaired cognitive function (assessed by the Glasgow Outcome Scale)
Identification of early predictors of adverse clinical outcome | 18 months
  Including clinical features and initial investigations which may be useful as a diagnostic tool.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Mason, MD, Principal Investigator — University of Sheffield

REFERENCES:
- [Background] Saab M, Gray A, Hodgkinson D, Irfan M. Warfarin and the apparent minor head injury. J Accid Emerg Med. 1996 May;13(3):208-9. doi: 10.1136/emj.13.3.208. PMID 8733663
- [Background] Stiell IG, Wells GA, Vandemheen K, Clement C, Lesiuk H, Laupacis A, McKnight RD, Verbeek R, Brison R, Cass D, Eisenhauer ME, Greenberg G, Worthington J. The Canadian CT Head Rule for patients with minor head injury. Lancet. 2001 May 5;357(9266):1391-6. doi: 10.1016/s0140-6736(00)04561-x. PMID 11356436
- [Background] Haydel MJ, Preston CA, Mills TJ, Luber S, Blaudeau E, DeBlieux PM. Indications for computed tomography in patients with minor head injury. N Engl J Med. 2000 Jul 13;343(2):100-5. doi: 10.1056/NEJM200007133430204. PMID 10891517
- [Background] Mower WR, Hoffman JR, Herbert M, Wolfson AB, Pollack CV Jr, Zucker MI; NEXUS II Investigators. National Emergency X-Radiography Utilization Study. Developing a clinical decision instrument to rule out intracranial injuries in patients with minor head trauma: methodology of the NEXUS II investigation. Ann Emerg Med. 2002 Nov;40(5):505-14. doi: 10.1067/mem.2002.129245. PMID 12399794
- [Background] Volans AP. The risks of minor head injury in the warfarinised patient. J Accid Emerg Med. 1998 May;15(3):159-61. doi: 10.1136/emj.15.3.159. PMID 9639176
- [Background] Hart RG, Boop BS, Anderson DC. Oral anticoagulants and intracranial hemorrhage. Facts and hypotheses. Stroke. 1995 Aug;26(8):1471-7. doi: 10.1161/01.str.26.8.1471. PMID 7631356
- [Background] Hylek EM, Singer DE. Risk factors for intracranial hemorrhage in outpatients taking warfarin. Ann Intern Med. 1994 Jun 1;120(11):897-902. doi: 10.7326/0003-4819-120-11-199406010-00001. PMID 8172435
- [Background] Ferrera PC, Bartfield JM. Outcomes of anticoagulated trauma patients. Am J Emerg Med. 1999 Mar;17(2):154-6. doi: 10.1016/s0735-6757(99)90050-5. PMID 10102316
- [Background] Mathiesen T, Benediktsdottir K, Johnsson H, Lindqvist M, von Holst H. Intracranial traumatic and non-traumatic haemorrhagic complications of warfarin treatment. Acta Neurol Scand. 1995 Mar;91(3):208-14. doi: 10.1111/j.1600-0404.1995.tb00436.x. PMID 7793238
- [Background] National Collaborating Centre for Acute Care (UK). Head Injury: Triage, Assessment, Investigation and Early Management of Head Injury in Infants, Children and Adults. London: National Collaborating Centre for Acute Care (UK); 2007 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK53036/ PMID 21563330
- [Background] Wilson JT, Pettigrew LE, Teasdale GM. Structured interviews for the Glasgow Outcome Scale and the extended Glasgow Outcome Scale: guidelines for their use. J Neurotrauma. 1998 Aug;15(8):573-85. doi: 10.1089/neu.1998.15.573. PMID 9726257
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Landefeld CS, Beyth RJ. Anticoagulant-related bleeding: clinical epidemiology, prediction, and prevention. Am J Med. 1993 Sep;95(3):315-28. doi: 10.1016/0002-9343(93)90285-w. PMID 8368229
- [Background] Fortuna GR, Mueller EW, James LE, Shutter LA, Butler KL. The impact of preinjury antiplatelet and anticoagulant pharmacotherapy on outcomes in elderly patients with hemorrhagic brain injury. Surgery. 2008 Oct;144(4):598-603; discussion 603-5. doi: 10.1016/j.surg.2008.06.009. Epub 2008 Aug 29. PMID 18847644
- [Background] Li J, Brown J, Levine M. Mild head injury, anticoagulants, and risk of intracranial injury. Lancet. 2001 Mar 10;357(9258):771-2. doi: 10.1016/S0140-6736(00)04163-5. PMID 11253975
- [Background] Gittleman AM, Ortiz AO, Keating DP, Katz DS. Indications for CT in patients receiving anticoagulation after head trauma. AJNR Am J Neuroradiol. 2005 Mar;26(3):603-6. PMID 15760873
- [Background] Lavoie A, Ratte S, Clas D, Demers J, Moore L, Martin M, Bergeron E. Preinjury warfarin use among elderly patients with closed head injuries in a trauma center. J Trauma. 2004 Apr;56(4):802-7. doi: 10.1097/01.ta.0000066183.02177.af. PMID 15187746
- [Background] Fabbri A, Vandelli A, Servadei F, Marchesini G. Coagulopathy and NICE recommendations for patients with mild head injury. J Neurol Neurosurg Psychiatry. 2004 Dec;75(12):1787-8. doi: 10.1136/jnnp.2004.041384. No abstract available. PMID 15548511
- [Background] Teasdale G, Murray G, Parker L, Jennett B. Adding up the Glasgow Coma Score. Acta Neurochir Suppl (Wien). 1979;28(1):13-6. doi: 10.1007/978-3-7091-4088-8_2. No abstract available. PMID 290137
- [Background] Fenwick E, Claxton K, Sculpher M. Representing uncertainty: the role of cost-effectiveness acceptability curves. Health Econ. 2001 Dec;10(8):779-87. doi: 10.1002/hec.635. PMID 11747057
- [Background] Felli JC, Hazen GB. Sensitivity analysis and the expected value of perfect information. Med Decis Making. 1998 Jan-Mar;18(1):95-109. doi: 10.1177/0272989X9801800117. PMID 9456214
- [Background] Ades AE, Lu G, Claxton K. Expected value of sample information calculations in medical decision modeling. Med Decis Making. 2004 Mar-Apr;24(2):207-27. doi: 10.1177/0272989X04263162. PMID 15090106
- [Background] Wilson JT, Edwards P, Fiddes H, Stewart E, Teasdale GM. Reliability of postal questionnaires for the Glasgow Outcome Scale. J Neurotrauma. 2002 Sep;19(9):999-1005. doi: 10.1089/089771502760341910. PMID 12482113
- [Derived] Mason S, Kuczawski M, Teare MD, Stevenson M, Goodacre S, Ramlakhan S, Morris F, Rothwell J. AHEAD Study: an observational study of the management of anticoagulated patients who suffer head injury. BMJ Open. 2017 Jan 13;7(1):e014324. doi: 10.1136/bmjopen-2016-014324. PMID 28087556
- [Derived] Kuczawski M, Stevenson M, Goodacre S, Teare MD, Ramlakhan S, Morris F, Mason S. Should all anticoagulated patients with head injury receive a CT scan? Decision-analysis modelling of an observational cohort. BMJ Open. 2016 Dec 13;6(12):e013742. doi: 10.1136/bmjopen-2016-013742. PMID 27974370